CLINICAL TRIAL: NCT03651921
Title: Co-creating and Testing the Reach and Effectiveness of an Integrated Peer-to-peer Self-management Program for Breast Cancer Survivors: a Pilot Study
Brief Title: Testing of the Cancer Thriving and Surviving Breast Cancer Program
Acronym: COSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuela Eicher (Other)
Collaborators: Swiss Cancer League (Other); Lindenhofgruppe AG (Industry)
Responsible Party: Sponsor-Investigator, Manuela Eicher, Associate Professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: ULausanne
Record Dates: First submitted 2018-05-01; First posted 2018-08-29 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Breast Neoplasm; Early-Stage Breast Cancer; Self-Management; Intervention; Cancer Survivorship
Keywords: Breast Cancer; Self-Management; Cancer Survivorship
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual follow-up care offered in the breast centers after primary treatment by breast care team (e. g. breast care nurses, gynaecologist, oncologist, psychologist).
- Usual care and CTS-BC-CH (Experimental): CTS-BC-CH as 7 weekly group session à 2.5 - 3 hours.
  Interventions: Behavioral: CTS-BC-CH

INTERVENTIONS:
Behavioral: CTS-BC-CH — CTS-BC-CH is a standardized program with 7 weekly group sessions (2.5. to 3 hours). The CTS-BC-CH focuses on building skills, sharing experiences, and support among the participants.
  Program elements are: Brainstorming, action plan formulation, action plan feedback, problem solving, and decision making.
  Arms: Usual care and CTS-BC-CH

SUMMARY:
The adjusted Cancer Thriving and Surviving Program (CTS) for women with breast cancer living in Switzerland (CTS-BC-CH) is a course of 7 weekly sessions of 2.5 - 3 hours led by trained peer-leaders (women with breast cancer experience). This pilot study aims to explore the reach of the CTS-BC-CH program (integrated into the clinical pathway) and to investigate its preliminary effectiveness with regard to Swiss breast cancer patients' self-efficacy and self-management.

DETAILED DESCRIPTION:
In 2016/17, the self-management program for cancer survivors, the Cancer Thriving and Surviving Program (CTS) was translated into German. The content of the CTS was adapted to breast cancer specific needs in three interdisciplinary workshops based on a participatory approach including active patient engagement. Additional disease-specific topics were developed and confirmed applying a multi-stakeholder e-rating approach. After a consensus meeting with the participation of breast cancer survivors, health care professional and international experts in the field of self-management, consensus on the program was reached in June 2017, resulting in the CTS-BC-CH program, i.e. a standardized manual for course leaders.

This pilot study aims to explore the reach of the CTS-BC-CH program (integrated into the clinical pathway) and to investigate its preliminary effectiveness for female Swiss breast cancer patients. The CTS-BC-CH is delivered in two breast cancer centers in in the German-speaking part of Switzerland as a group-based program with seven weekly sessions of 2.5 - 3 hours led by trained peer-leaders. Course leaders have to complete a 4-days training provided by certified master trainers. First, participants are enrolled for usual care, followed by participants who will attend the CTS-BC-CH course. Participants will complete self-reported questionnaires at three time points over a period of 6 months.

ELIGIBILITY:
Inclusion breast cancer patients

* female gender
* written informed consent
* aged 18 years or older
* diagnosed with an early stage breast cancer (stage 0, stage I, stage IIA, stage IIB, and stage IIIA breast cancers)
* completed primary therapy (i. e. surgery, chemotherapy and/or radiation therapy)
* at the beginning of follow-up care (including long-term endocrine therapy or targeted therapy)
* free of recurrence
* mentally able to participate, assessment of the psychological state performed by the responsible psychologist/psycho-oncologist in the breast center
* treated in the participating breast center

Inclusion course leaders

* female gender
* written informed consent
* aged 18 years or older
* diagnosed with an early stage breast cancer (stage 0, stage I, stage IIA, stage IIB, and stage IIIA breast cancers)
* > than 2 years post diagnosis
* free of recurrence
* mentally able to participate, assessment of the psychological state performed by the responsible psychologist/psycho-oncologist in the breast center
* treated in the participating breast center
* willing to participate in a course leaders training

Exclusion breast cancer patients and course leaders

* participation in another psycho-social intervention study
* known illiteracy (reading and writing difficulties)
* lack of language proficiency (German)

Inclusion breast care nurses for CTS-BC-CH implementation

* female gender
* employed at breast care center > 1 year
* participation in 4-days CTS-BC-CH course leader training

Inclusion breast care nurses for evaluating self-management support practices

* nurses: graduated with a nurses diploma > 1 year of breast cancer care experience

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female breast cancer patients or female breast care nurses.
Enrollment: 39 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Reach of intervention assessed by ratio of eligible patients vs. participating patients | 21 weeks after baseline
Changes in self-management skills assessed by heiQ | Change from baseline to 20 weeks after baseline
  Assessed by the Health Education Impact Questionnaire (heiQ)

SECONDARY OUTCOMES:
Change in patient-reported self-efficacy assessed by SES6G | Change from baseline to 20 weeks after baseline
  Assessed by the Self-Efficacy for Managing Chronic Disease Scale (SES6G)
Change in patient-reported health literacy assessed by HLS-EU-Q6 | Change from baseline to 20 weeks after baseline
  Assessed by the Health Literacy Scale Europe (HLS-EU-Q6)
Change in patient-reported symptom burden assessed by BCPT Symptom Scales | Change from baseline to 20 weeks after baseline
  Assessed by the Breast Cancer Prevention Trial (BCPT) Symptom Scales
Change in patient-reported health service navigation assessed by heiQ | Change from baseline to 20 weeks after baseline
  Assessed by a subscale of the Health Education Impact Questionnaire (heiQ)
Change in nurse-reported self-efficacy and self-management support practices assessed by SEPSS | Change from baseline to 30 weeks after baseline
  Assessed by the Self-Efficacy and Performance in Self-management Support (SEPSS) measure

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Eicher, Prof. Dr., Study Director — Institute of Higher Education and Reserach in Health Care - IUFRS University of Lausanne and University Hospital of Lausanne; Joerg Haselbeck, Dr., Study Director — Swiss Cancer League Berne; Formely: Careum Stiftung, Kompetenzzentrum Patientenbildung; Karin Ribi, Dr. phil., Study Chair — International Breast Cancer Study Group (IBCSG); Corinne Urech, Dr. phil., Study Chair — University Hospital, Basel, Switzerland; Karin Holm, Study Chair — Patient Advocats for Cancer Reserach and Treamtment (Association PARCT)
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Inselspital Bern, Bern

IPD SHARING:
Plan to Share IPD: Undecided